CLINICAL TRIAL: NCT00023686
Title: A Randomized Trial of Radical Prostatectomy Versus Brachytherapy for Patients With T1c or T2a N0 M0 Prostate Cancer
Brief Title: Surgery Versus Internal Radiation in Treating Patients With Stage II Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACOSOG-Z0070; ACOSOG-Z0070; CDR0000068851 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surgical Procedures, Operative; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- surgery (Experimental): Patients undergo radical prostatectomy.
  Patients are followed every 6 months for 5 years and then annually thereafter.
  Interventions: Procedure: surgery
- radiation (Experimental): Patients undergo brachytherapy with implanted iodine I 125 or palladium Pd 103 seeds.
  Patients are followed every 6 months for 5 years and then annually thereafter.
  Interventions: Radiation: radiation

INTERVENTIONS:
Procedure: surgery
  Arms: surgery
Radiation: radiation
  Arms: radiation

SUMMARY:
RATIONALE: Internal radiation uses radioactive material placed directly into or near a tumor to kill tumor cells. It is not yet known whether surgery is more effective than internal radiation in treating prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of surgery with that of internal radiation in treating patients who have stage II prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare overall survival in patients with stage II prostate cancer treated with radical prostatectomy vs brachytherapy.
* Compare metastasis-free survival and probability of survival without symptoms of patients treated with these regimens.
* Compare the side effects of these treatment regimens in these patients.

OUTLINE: This is a randomized study. Patients are randomized to one of two treatment arms.

* Arm I: Patients undergo radical prostatectomy.
* Arm II: Patients undergo brachytherapy with implanted iodine I 125 or palladium Pd 103 seeds Patients are followed every 6 months for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 1,980 patients (990 per treatment arm) will be accrued for this study within 5.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate within the past 120 days

  * T1c-T2a, N0, M0
* No bilateral disease
* Prostate-specific antigen (PSA) no greater than 10 ng/mL

  * In patients with prior neoadjuvant hormonal therapy (NHT), PSA must be less than 10 ng/mL prior to therapy
* Gleason score no greater than 6
* Prostate gland less than 60 cc on transrectal ultrasound or with minimal pubic arch interference OR
* Prostate gland 60 cc or greater prior to NHT allowed if prostate size has been reduced to less than 60 cc by NHT

PATIENT CHARACTERISTICS:

Age:

* 75 and under

Performance status:

* ECOG 0-2 OR
* Zubrod 0-2

Renal:

* Creatinine no greater than 3 mg/dL

Cardiovascular:

* No significant cardiovascular disease
* No New York Heart Association class III or IV heart disease

Other:

* No other malignancy within the past 5 years except effectively treated basal cell or squamous cell skin cancer or other malignancy at low risk for recurrence
* No other condition that would preclude study

PRIOR CONCURRENT THERAPY:

Endocrine therapy:

* See Disease Characteristics
* At least 90 days since prior NHT

  * Duration of therapy no greater than 120 days
* No concurrent NHT

Radiotherapy:

* No prior radiotherapy to pelvis

Surgery:

* No prior surgery for prostate cancer or benign disease, including:

  * Transurethral resection of the prostate
  * Transurethral resection of the bladder neck
  * Cryotherapy
  * Laser ablation
  * Microwave therapy

Max Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2001-10; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
overall survival | Up to 10 years

SECONDARY OUTCOMES:
disease free survival | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul H. Lange, MD, Study Chair — University of Washington
Locations (36):
- United States (30):
  - St. Vincent Cancer Center, Little Rock, Arkansas
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Kansas Cancer Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Northeast Heights Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Wellspan Health - York Cancer Center, York, Pennsylvania
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - American Fork Hospital, American Fork, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Fletcher Allen Health Care - Medical Center Campus, Burlington, Vermont
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington
- Canada (6):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec

REFERENCES:
- [Background] Crook J, Wallace K, Jewett M, et al.: Enhancing enrollment in difficult randomized trials: the profile of men accepting randomization to SPIRIT (surgical prostatectomy vs interstitial radiation). [Abstract] 2006 Prostate Cancer Symposium, February 24-26, 2006, San Francisco, CA. A-295, 2006.
- [Background] Wallace K, Fleshner N, Jewett M, Basiuk J, Crook J. Impact of a multi-disciplinary patient education session on accrual to a difficult clinical trial: the Toronto experience with the surgical prostatectomy versus interstitial radiation intervention trial. J Clin Oncol. 2006 Sep 1;24(25):4158-62. doi: 10.1200/JCO.2006.06.3875. PMID 16943531
- [Result] Crook JM, Gomez-Iturriaga A, Wallace K, Ma C, Fung S, Alibhai S, Jewett M, Fleshner N. Comparison of health-related quality of life 5 years after SPIRIT: Surgical Prostatectomy Versus Interstitial Radiation Intervention Trial. J Clin Oncol. 2011 Feb 1;29(4):362-8. doi: 10.1200/JCO.2010.31.7305. Epub 2010 Dec 13. PMID 21149658
- [Result] Crook JM, Gomez-Iturriaga A, Wallace K, et al.: Comparison of health-related quality of life 5 years after SPIRIT (Surgical Prostatectomy [RP] versus Interstitial Radiation [BT] Intervention trial ACOSOG Z0070). [Abstract] 2010 Genitourinary Cancers Symposium, March 5-7, 2010, San Francisco, California. A-11, 2010.